CLINICAL TRIAL: NCT03666455
Title: Treating Pain With Acceptance and Commitment Therapy Trial
Acronym: T-PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: University of Kansas Medical Center (Other); University of North Carolina, Chapel Hill (Other); University of Kentucky (Other)
Responsible Party: Principal Investigator, Robert L Rhyne, Professor & Vice Chair of Research, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-270
Record Dates: First submitted 2018-07-20; First posted 2018-09-11 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Acceptance and Commitment Therapy; Chronic Pain; Opioid Use
MeSH Terms: conditions — Chronic Pain | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Study Design: Mixed methods, intervention trial, feasibility study, with sequential and concurrent quantitative and qualitative data collection before, during, and after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acceptance and Commitment Therapy (Experimental): The intervention consists of eight individual (one-on-one) acceptance and commitment therapy sessions approximately one week apart over a 12-week period.
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Acceptance and commitment therapy (ACT) is a type of psychotherapy, or cognitive behavioral therapy, that aims to help patients focus on the present, accept their situation, and find positive coping skills.

SUMMARY:
The long-term goal is to define best practices for diminishing the risk of high opioid doses used to treat chronic non-cancer pain (CNCP) patients while optimizing pain outcomes and functional levels of activity, emotional functioning, and quality of life. The short-term goal is to assess the feasibility of multiple Clinical and Translational Research Award (CTSA) sites working together to perform and study the effects of a cognitive behavioral therapy intervention in a future randomized controlled trial (RCT) among CNCP patients in rural primary care practices in each CTSA state.

DETAILED DESCRIPTION:
The long-term goal is to define best practices for diminishing the risk of high opioid doses used to treat chronic non-cancer pain (CNCP) patients while optimizing pain outcomes and functional levels of activity, emotional functioning, and quality of life. The short-term goal is to assess the feasibility of multiple Clinical and Translational Research Award (CTSA) sites working together to perform and study the effects of a cognitive behavioral therapy intervention in a future randomized controlled trial (RCT) among CNCP patients in rural primary care practices in each CTSA state.

The current feasibility study uses a multi-site, pragmatic, community-based, mixed methods design to assess the feasibility of multiple CTSA locations working together to administer the evidence-based intervention, Acceptance and Commitment Therapy (ACT), to reduce harmful opioid use among CNCP patients. This mixed methods study will have a quantitative arm and a qualitative arm. Following this feasibility study, the team will use the resulting preliminary data to apply for a larger grant to implement a larger multi-site RCT at the same sites.

The specific aims of this feasibility study are:

1. To conduct a multi-site, mixed methods study to demonstrate the feasibility of performing a future pragmatic RCT on the effectiveness of treating CNCP with Acceptance and Commitment Therapy (ACT), delivered in rural primary healthcare practices, with the goal of decreasing chronic, harmful opioid use among rural populations.
2. To generate preliminary data that will be used to apply for a larger multi-site RCT study that would test the effectiveness of ACT in the same population of rural pain patients.

The feasibility study hypothesis is that the study team can demonstrate the ability for multiple CTSA sites to work together on a small research project in rural primary care practices, among rural patients with chronic non-cancer pain on long-term opioid therapy. The team will show that it is feasible to implement the intervention ACT in a future larger RCT study, which would test its effectiveness at reducing or eliminating opioid use while managing chronic pain.

The hypothesis for preliminary data collection and a larger RCT is that ACT, which has been shown to be an effective treatment for chronic pain, will be effective at reducing or eliminating opioid use for CNCP patients in rural primary care practices.

Research questions:

1. Quantitative research questions: Is ACT delivered in a rural primary care practices an effective alternative to opioids in managing chronic pain? How does ACT impact chronic pain in rural primary healthcare patients?
2. Qualitative research question: How do participants evaluate ACT as an alternative to opioids in their pain management?

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (21-65 years of age).
* Has a diagnosis of CNCP (> 3 months). We will limit the diagnostic inclusion criteria to the most common pain diagnoses (excluding headache): low back, multi-site/full body (e.g., fibromyalgia, and various kinds of arthritis), neck, lower extremity, and abdomen.
* Being prescribed chronic opioid medications for the pain.
* Mentally and physically able to participate in data collection (namely, completing an extensive survey at three points in time, attending 8 one-hour therapy sessions, and participating in an interview by the research staff).

Exclusion Criteria:

* Children under the age of 21 will be excluded from participating because this study is examining ACT in adults with CNCP. Pregnant women will be excluded because their use of opioids presents a special therapeutic circumstance out of the scope of this study. People who are not fluent in English will be excluded because this is a small feasibility study and we do not have the resources to conduct the intervention or collect data in other languages.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Primary study outcome will be the Success Scale of the Chronic Pain Values Inventory. | One year
  Primary study outcome will be the Success Scale of the Chronic Pain Values Inventory (CPVI). Based on an in-progress meta-analysis of unidisciplinary Acceptance and Commitment Therapy for chronic pain, we expect a post-treatment effect size of d = .80 (95% CI: .41 - 1.20).
  Construct: The CPVI has 12 items that measure, "which values are important to an individual and to assess the degree of success they are having in following their values" and "has supported its use in a contextual analysis of pain and as part of a treatment for chronic pain." Scale ranges: 0 to 5. First sore is mean success rating; second score is mean discrepancy rating. Outcome measures: "Low success in living in accordance to an important value is presumed to entail greater suffering than low success in living in accordance to a value that is relatively unimportant."

SECONDARY OUTCOMES:
The secondary study outcome will be the Pain Interference Scale of the Brief Pain Inventory. | One year
  The secondary study outcome will be the Pain Interference Scale of the Brief Pain Inventory (BPI). Based on an in-progress meta-analysis of unidisciplinary Acceptance and Commitment Therapy for chronic pain, we expect a post-treatment effect size of d = .40 (95% CI: .17 - .64).
  Construct: The BPI measures chronic cancer- and noncancer-related pain. Scale ranges: Scale of 0 to 10; patients rate current pain intensity, pain in the last 24 hours, and pain interference in quality of life. Higher scores equal greater pain and/or greater interference. Outcome measures: A decrease in scores over time indicates an improvement of pain and less interference of pain on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rhyne, MD, Principal Investigator — University of New Mexico
Locations (4):
- United States (4):
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - University of New Mexico, Albuquerque, New Mexico
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tan G, Jensen MP, Thornby JI, Shanti BF. Validation of the Brief Pain Inventory for chronic nonmalignant pain. J Pain. 2004 Mar;5(2):133-7. doi: 10.1016/j.jpain.2003.12.005. PMID 15042521
- [Background] Keller S, Bann CM, Dodd SL, Schein J, Mendoza TR, Cleeland CS. Validity of the brief pain inventory for use in documenting the outcomes of patients with noncancer pain. Clin J Pain. 2004 Sep-Oct;20(5):309-18. doi: 10.1097/00002508-200409000-00005. PMID 15322437
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] McCracken LM, Yang SY. The role of values in a contextual cognitive-behavioral approach to chronic pain. Pain. 2006 Jul;123(1-2):137-45. doi: 10.1016/j.pain.2006.02.021. Epub 2006 Mar 29. PMID 16564627